CLINICAL TRIAL: NCT04812145
Title: Role of Hypofractionated Radiotherapy With Concurrent Gemcitabine in Treatment of Urinary Bladder Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mostafa Abdelzaher Mohamed, Principal Investigator, Assiut University
Other Study IDs: U.Bladder Cancer Radiotherapy
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Chemoradiation — Hypofractionated radiotherapy with concurrent Gemcitabine

SUMMARY:
Estimate the response to modified hypofractionated radiotherapy concurrent with Gemcitabine in urinary bladder cancer patients .

Estimate local control, relapse free survival, overall survival and bladder preservation rate. Evaluate the toxicity of a modified hypofractionated chemoradiotherapy protocol for patients with invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

- Pathologically confirmation of transitional cell carcinoma . Non metastatic invasive bladder cancer (TNM0) Any age group ≥ 18 years. Non pregnant female patients.

Exclusion Criteria:

- Other pathology than Transitional cell carcinoma Metastatic Patient Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urinary bladder cancer patient histologically proved Transitional cell carcinoma received concurrent chemoradiation with gemcaitabine
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Response to hypofractionated radiotherapy concurrent with Gemcitabine in urinary bladder cancer | baseline
  Estimate Disease free survival .

REFERENCES:
- [Background] 1. Siegel, R.L., K.D. Miller, and A. Jemal, Cancer statistics, 2019. CA: a cancer journal for clinicians, 2019. 69(1): p. 7-34. 2. Staerkel,Ro, J.Y., G.A. andAyala, A.G. Cytologic and histologic features of superficial bladder cancer. The Urologic clinics of North America, 1992. 19(3): p. 435-453. 3. Witjes, J.A., T. Lebret, E.M. Compérat, N.C. Cowan, M. De Santis, H.M. Bruins, et al., Updated 2016 EAU guidelines on muscle-invasive and metastatic bladder cancer. European urology, 2017. 71(3): p. 462-475. 4. De Santis, M. Bachner , M. Cerveny, et al. Combined chemoradiotherapy with gemcitabine in patients with locally advanced inoperable transitional cell carcinoma of the urinary bladder and/or in patients ineligible for surgery: a phase I trial. Ann Oncol, 25 (2014), pp. 1789-1794. 5. Kimura, T., H. Ishikawa, T. Kojima, S. Kandori, T. Kawahara, Y. Sekino, et al., Bladder preservation therapy for muscle invasive bladder cancer: the past, present and future. Japanese Journal of Clinical Oncology, 2020. 50(10): p. 1097-1107. 6. Flaig, T.W., P.E. Spiess, N. Agarwal, R. Bangs, S.A. Boorjian, M.K. Buyyounouski, et al., NCCN guidelines insights: bladder cancer, version 5.2018. Journal of the National Comprehensive Cancer Network, 2018. 16(9): p. 1041-1053. 7. Mitin, T., A. George, A.L. Zietman, N.M. Heney, D.S. Kaufman, R.G. Uzzo, et al., Long-term outcomes among patients who achieve complete or near-complete responses after the induction phase of bladder-preserving combined-modality therapy for muscle-invasive bladder cancer: a pooled analysis of NRG Oncology/RTOG 9906 and 0233. International Journal of Radiation Oncology* Biology* Physics, 2016. 94(1): p. 67-74. 8. Mak, K.S., A.B. Smith, A. Eidelman, R. Clayman, A. Niemierko, J.-S. Cheng, et al., Quality of life in long-term survivors of muscle-invasive bladder cancer. International Journal of Radiation Oncology* Biology* Physics, 2016. 96(5): p. 1028-1036. 9. Azria, D., O. Riou, X. Rebillard, S. Thezenas, R. Thuret, P. Fenoglietto, et al., Combined chemoradiation therapy with twice-weekly gemcitabine and cisplatin for organ preservation in muscle-invasive bladder cancer: long-term results of a phase 1 trial. International Journal of Radiation Oncology* Biology* Physics, 2014. 88(4): p. 853-859. 10. Shipley, W.U., G.R. Prout, A.B. Einstein, L.J. Coombs, Z. Wajsman, M.S. Soloway, et al., Treatment of invasive bladder cancer by cisplatin and radiation in patients unsuited for surgery. Jama, 1987. 258(7): p. 931-935. 11. Borut K, Lijana ZK. Phase I study of radiochemothearpy with gemcitabine in invasive bladder cancer. RadiotherOncol 2012;102:412-5.